CLINICAL TRIAL: NCT03584308
Title: Efficacy and Safety of VIUSID® Plus GLIZIGEN® in Patients With Papilloma Virus Esophageal. Phase II Clinical Trial
Brief Title: Efficacy of VIUSID® Plus GLIZIGEN® in Patients With Papilloma Virus Esophageal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIUSID-GLIZ-PAPILOMA
Record Dates: First submitted 2018-06-28; First posted 2018-07-12 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2018-06

CONDITIONS: Papilloma Viral Infection; Papillomavirus Infections; Esophageal Viral Wart; Esophageal Verrucous Carcinoma
Keywords: Papillomavirus; Viusid; Glizigen; Papilloma virus Esophageal; Antioxidant
MeSH Terms: conditions — Papillomavirus Infections | interventions — Viusid

STUDY DESIGN:
Intervention Model Description: Random assignment, through a list obtained by computer. Patients will be randomized in the consultation of the upper digestive tract, once the anatomopathological result with the presence of coilocytes is received, and they meet the established selection criteria.
Who Masked: Participant, Investigator
Masking Description: A double blind. To achieve the masking of the research product, these have been labeled by a computerized randomized balanced list, which will be in the possession of the promoter and the study Biostatistician. The masking will be maintained until the analysis of the data. However, access to the code will be allowed if serious adverse events arise related to the research product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Viusid® + Glizigen® (Experimental): The experimental arm will receive nutritional supplements Viusid + Glizigen
  Interventions: Dietary Supplement: Viusid®; Dietary Supplement: Glizigen®
- Placebo (Placebo Comparator): The control group will receive a placebo of both (Viusid and Glizigen).
  Interventions: Dietary Supplement: Viusid Placebo; Dietary Supplement: Glizigen Placebo

INTERVENTIONS:
Dietary Supplement: Viusid® — The VIUSID nutritional supplement is presented in the form of envelopes and will be administered orally diluted in water, juice or milk, according to the patient's preference and will be administered 3 times a day, 15 minutes before breakfast, lunch and dinner.
  Arms: Viusid® + Glizigen®
Dietary Supplement: Glizigen® — The GLIZIGEN® product is presented in spray bottles and will be administered orally to swallow, away from meals 2 times a day.
  Arms: Viusid® + Glizigen®
Dietary Supplement: Viusid Placebo — The placebo of VIUSID nutritional supplement is presented in the form of envelopes and will be administered orally diluted in water, juice or milk, according to the patient's preference and will be administered 3 times a day, 15 minutes before breakfast, lunch and dinner .
  Arms: Placebo
Dietary Supplement: Glizigen Placebo — The placebo of GLIZIGEN® product is presented in spray bottles and will be administered orally to swallow, away from meals 2 times a day.
  Arms: Placebo

SUMMARY:
A randomized, double-blind, phase II clinical trial was conducted versus placebo in 110 patients with esophageal human papillomavirus. The experimental group will receive the VIUSID® plus GLIZIGEN® nutritional supplements, administered on an outpatient basis for 3 months. The control group will receive placebo from Viusid plus Glizigen placebo. It is expected that patients in the experimental group have a 30% higher rate of elimination of the virus than patients in the placebo group after treatment. The study will be conducted in the Superior Digestive Tract consultation of the Institute of Gastroenterology of Havana, Cuba.

DETAILED DESCRIPTION:
Initially the study was planned as an adaptive study without seams, phase II / III for 150 patients. 75 in each therapeutic arm. The sample size was calculated with parameters of phase III studies, but establishing an early stop rule, with an intermediate analysis. For the calculation it was taken into account that the expected percentage of elimination of the virus by spontaneous remission in immunocompetent patients, reported internationally is on average 35%. It is intended that in the group of patients to whom VIUSID® plus GLIZIGEN® will be administered, this figure is ≥ 65%. In other words, it is desired to reach a minimum difference of approximately 30% between both groups. Considering a type I error of 5% (adjusted to 2.5% by an intermediate evaluation), a power of 90%, plus 5% of dropouts or losses to follow-up, the minimum number of patients to recruit is 150 patients in total , 75 in each therapeutic arm.

However, by decision of the promoter the study was stopped with 55 patients in each arm, 110 patients in total. And established as a phase II trial.

ELIGIBILITY:
Inclusion Criteria:

* Older adults between 18 and 65 years of both sexes.
* Patients residing in the provinces of Havana, Artemisa and Mayabeque.
* Voluntariness of the patient to participate in the study. Informed and written consent.
* Women of childbearing age should have negative pregnancy test or use effective contraceptive methods such as intrauterine devices, hormonal contraceptives, barrier method or tubal ligation.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Contraindication to the performance of upper digestive endoscopy.
* Psychiatric conditions that do not favor the administration of treatment and follow-up.
* History of hypersensitivity to another similar product.
* Severe acute allergic states.
* Patients with concomitant diagnosis of esophageal tumor or other causes of infectious esophagitis.
* Present an associated chronic illness in the decompensation phase (heart disease, diabetes, hypertension, renal failure, AIDSl).
* Patients who are receiving another product under investigation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of the lesions of the virus in esophageal mucosal tissue sample | 3 months
  Absence of coilocytes / papilloma in the paraffin sample
Clinical negativization of the virus in esophageal mucosal tissue sample | 3 months
  Negativization of the virus in fresh sample of the mucosa in the PCR study

SECONDARY OUTCOMES:
Evaluation of esophageal pathology | 3 months
  Acanthosis: Yes or No
Evaluation of esophageal pathology | 3 months
  Papillary hyperplasia lamina propria: Yes or no
Evaluation of esophageal pathology | 3 months
  Hyperplasia of the basal layer of the epithelium: Yes or No
Evaluation of esophageal pathology | 3 months
  Dyskeratosis: Yes or No
Evaluation of esophageal pathology | 3 months
  Dysplasia: Yes (Low Degree or High Degree) or No
Toxicity due to the Treatment administered | 3 months
  It will be determined through the reporting of adverse events that are presented to the research product

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Institute, Vedado, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR